CLINICAL TRIAL: NCT03662763
Title: Phase 3,Double Blind,Placebo-controlled,Multicentre,Randomised-withdrawal,Long-term Maintenance of Efficacy&Safety Study of Extended-release Guanfacine Hydrochloride in Children/Adolescents Aged 6-17 With ADHD
Brief Title: Extended-release Guanfacine Hydrochloride in Children/Adolescents With Attention-deficit/Hyperactivity
Acronym: SPD503-315
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101081
Record Dates: First submitted 2011-08-09; First posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Attention Deficit Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule
- Extended-release Guanfacine Hydrochloride (SPD503) (Experimental)
  Interventions: Drug: Extended-release Guanfacine Hydrochloride (SPD503)

INTERVENTIONS:
Drug: Extended-release Guanfacine Hydrochloride (SPD503) — dosing in all subjects will initiate with 1mg/day, and may be increased by 1 mg increments after a minimum of 1 week on the current dose to the maximum doses based on age and weight.
  Other Names: Extended-release Guanfacine Hydrochloride; SPD503
  Arms: Extended-release Guanfacine Hydrochloride (SPD503)
Drug: Placebo oral capsule
  Arms: Placebo

SUMMARY:
A study to evaluate the long term maintenance of efficacy of using Guanfacine Hydrochloride (SPD-503) for the treatment of ADHD in Children aged 6-17 years in Europe, Australia, Canada and the US.

DETAILED DESCRIPTION:
The SPD503-315 clinical program has studied the efficacy, safety, and tolerability of this product in treating symptoms of ADHD in children and adolescents aged 6-17 through short-term, placebo-controlled studies and long-termn, open-label studies. This study will more rigorously assess the long-term maintenance of efficacy using a placebo-controlled, randomised-withdrawal design. To date, all of the completed studies conducted as part of the SPD503 proigram have enrolled subjects from the US. This study is designed to evaluate the long-term maintenance of efficacy of SPD503 for the treatment of ADHD in children aged 6-17 years in Europe, Australia, Canada and US.

ELIGIBILITY:
Inclusion Criteria:

* male or female, aged 6-17 years at the time of consent/assent at Screening/Visit 1
* subject meets DSM-IV-TR criteria for primaru diagnosis of ADHD
* subject has a minimum ADHD-RS-IV total score of 32 at enrolment/visit 2
* subject has a minimum CGI-S score of 4 at Enrolment/Visit 2
* subject is able to swallow intact tablets

Exclusion Criteria:

* subject has a current controlled or uncontrolled, co-morbid psychiatric diagnosis.
* subject has a know history or presence of structural cardiac abnormalities
* subject with orthostatic hyupotension or a known history of controlled or uncontrolled hypertension
* current use of any prohibited medication or other medications, including herbal supplements that affet blood pressure, or heart rate or that have CNS effects or affect cognitive performance
* subject is significant overweight based on Centre for disease control and prevention BMI for age gender specific charts. Significantly overweight is defined as a BMI >95 th percentile Children aged 6-12 years with a body weight ,25,0kg, or adolescents aged 13-17 years with a body weight <43 kg or >91 kg at screening/visit 1
* subject is currently considered a suicide risk in the opinion of the investigator
* history of failure to respond to an adequate trial of an alfa2-agonist for the treatment of ADHD.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Attention Deficit Hyperactivity Disorder-Rating Scale -IV | 13 weeks

SECONDARY OUTCOMES:
Clinical Global Impressions-Severity score | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andries Korebrits, prof. Dr., Principal Investigator — psychiatrie
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands